CLINICAL TRIAL: NCT04281017
Title: Effect of Position and Anesthetic Choice in Intraocular Pressure in Robotic GYN (Gynecologic) Oncology Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB202000034; OCR33027 (Other: University of Florida)
Record Dates: First submitted 2020-02-20; First posted 2020-02-21 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Intraocular Pressure; Oncology
Keywords: robotic gynecologic surgery
MeSH Terms: conditions — Neoplasms | interventions — Balanced Anesthesia

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TIVA anesthesia (Experimental): Induction with 1% propofol (2-3 mg/kg), fentanyl (1-3 mg/kg), and Rocuronium 1-1.5 mg/kg. Before the injection of propofol, 5 mL 1% lidocaine (50 mg) to limit any discomfort caused by the propofol injection. After endotracheal intubation, intravenous infusion of propofol, lidocaine, ketamine or narcotic as deemed appropriate by anesthesiologist. There will be no inhalation anesthetic used. Ventilation with oxygen and air mixture (50%/50%) and titrated to keep the mean arterial pressure within 20% of its preinduction value. Muscle relaxation maintain using Aliquots of rocuronium to 0 to 1 train-of-4 twitch response of adductor pollicis. During surgery, mechanical ventilation using pressure-controlled mode (peak inspiratory pressure 30 cm H2O). We aim for Tidal volume of 5-7 ml/Kg of ideal body weight with a positive end-expiratory pressure of 5 cm H2O, and a respiratory rate to maintain end-tidal carbon dioxide between 30 to 40 mm Hg.
  Interventions: Drug: TIVA
- Balanced anesthesia (Active Comparator): Induction with 1% propofol (2-3 mg/kg), fentanyl (1-3 mg/kg), and Rocuronium 1-1.5 mg/kg. Before the injection of propofol, 5 mL 1% lidocaine (50 mg) to limit any discomfort caused by the propofol injection. After endotracheal intubation, the depth of anesthesia will be maintained at a minimum alveolar concentration of 1 to 1.25 using isoflurane in oxygen and air mixture (50%/50%) and titrated to keep the mean arterial pressure within 20% of its preinduction value. Muscle relaxation maintain using Aliquots of rocuronium to 0 to 1 train-of-4 twitch response of adductor pollicis. During the surgery, subjects will be mechanically ventilated using pressure-controlled mode (peak inspiratory pressure 30 cm H2O). We aim for Tidal volume of 5-7 ml/Kg of ideal body weight with a positive end-expiratory pressure of 5 cm H2O, and a respiratory rate to maintain end-tidal carbon dioxide between 30 to 40 mm Hg.
  Interventions: Drug: Balanced anesthesia

INTERVENTIONS:
Drug: TIVA — Induction with 1% propofol (2-3 mg/kg), fentanyl (1-3 mg/kg), and Rocuronium 1-1.5 mg/kg. Before the injection of propofol, 5 mL 1% lidocaine (50 mg)
  Arms: TIVA anesthesia
Drug: Balanced anesthesia — Induction with 1% propofol (2-3 mg/kg), fentanyl (1-3 mg/kg), and Rocuronium 1-1.5 mg/kg. Before the injection of propofol, 5 mL 1% lidocaine (50 mg
  Arms: Balanced anesthesia

SUMMARY:
Steep Trendelenburg positioning and insufflation of the abdominal cavity have shown to increase intra ocular pressure. Different anesthetic techniques can alter intra ocular pressure and a small pilot study showed decrease in Intraocular Pressure (IOP) in robotic case in steep Trendelenburg with IV anesthetics (TIVA).

We want to quantify the degree of change in Intraocular Pressure (IOP) in female patients undergoing robotic procedures for cancer. We want to detect the difference in increase of pressure with total IV anesthesia versus conventional balanced anesthesia

DETAILED DESCRIPTION:
During the day of surgery, the anesthesiologist trained by an ophthalmologist, will measure each eye's Intraocular Pressure (IOP) using a tonometer for both the Trendelenburg with IV anesthetics (TIVA) and propofol/fentanyl/rocuronium arms of the study. (The Tono-Pen XL Medtronic Solan, Jacksonville, FL) The Intraocular Pressure (IOP) for both eyes will be measured at seven time points:

Time 1 induction after administration of sedative and local anesthesia in the eye. Both eyes of the patient will anesthetized using topical proparacaine hydrochloride ophthalmic solution 0.5%.

Time 2 Post induction table 0 degrees Time 3 Supine after pneumoperitoneum with 14 mmHg pressure Time 4 After docking robot at correct Trendelenburg positioned measured by a level Time 5 After undocking and before moving supine Time 6 Supine and before extubation. If the intraocular pressure remains elevated above 19 mmHg will require a 7th measurement in PACU with HOB at 30 degrees and if the pressure still at or above 19 ophthalmology consult initiated.

Time 7 if needed, see above

If the patient has any increased reading at the end of the procedure, the same attending anesthesiologist in the post-operative recovery area prior to discharge will do a post op measurement. Any abnormal readings will prompt an ophthalmology consult and follow up with ophthalmology department.

ELIGIBILITY:
Inclusion Criteria:

* Females ≥ eighteen years of age
* Written informed consent obtained from the subject and the subject agrees to comply with all the study-related procedures
* Subjects must be planning to receive robotic surgery for gynecological cancer or high suspicion of cancer (these subject will be withdrawn if it his proven they don't have cancer)
* Subjects must be cleared for surgery by the pre-anesthesia clinic
* All robotic GYN cancer patients 18 years of age and older with any preexisting medical conditions that are deemed ready for surgery by the pre anesthesia clinic

Exclusion Criteria:

* Known increased intraocular pressure, prior eye surgery within a month, eye conditions where the ophthalmologist would not allow an intra ocular pressure measurement
* Subjects with a previous treatment of diagnosis of increased intraocular pressure
* Subjects who have undergone eye surgery in the 30 days prior to consent
* Subjects for whom an ophthalmologist has determined cannot undergo intraocular pressure measurement

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — GYN cases only done in female subjects
Enrollment: 40 (Estimated)
Dates: Start 2020-11-10 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2027-06-18 (Estimated)

PRIMARY OUTCOMES:
Quantify the degree of change in intra ocular pressure in female patients undergoing robotic procedures | Day of Surgery
  quantify the degree of change in IOP in female patients undergoing robotic procedures for cancer

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Mehta, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No